CLINICAL TRIAL: NCT02169154
Title: A Cumulative Skin Irritation Study Investigating the Skin Irritancy Potential of MFC51123 Diclofenac-Menthol Gel
Brief Title: A Safety Study to Investigate the Skin Irritancy Potential of Diclofenac-Menthol Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 202187; RH02170 (Other: GSK)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diclofenac; Menthol; Sodium Dodecyl Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Diclofenac Sodium/Menthol Gel (Experimental): 1% diclofenac sodium + 3% menthol
  Interventions: Drug: 1% Diclofenac Sodium; Drug: 3% Menthol
- Diclofenac Gel (Active Comparator): 1% diclofenac sodium + 0.09% menthol
  Interventions: Drug: 1% Diclofenac Sodium; Drug: 0.09% Menthol
- Menthol Gel (Active Comparator): 3% menthol
  Interventions: Drug: 3% Menthol
- Placebo Gel (Placebo Comparator): 0.09% menthol
  Interventions: Drug: 0.09% Menthol
- Voltaren Gel (Active Comparator): 1% diclofenac sodium
  Interventions: Drug: 1% Diclofenac Sodium
- Sodium lauryl sulfate (Placebo Comparator): 0.2% Sodium lauryl sulfate
  Interventions: Drug: 0.2% Sodium Lauryl Sulfate
- Saline (Placebo Comparator): 0.9% saline
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: 1% Diclofenac Sodium — 1% diclofenac sodium
  Arms: Diclofenac Gel; Diclofenac Sodium/Menthol Gel; Voltaren Gel
Drug: 3% Menthol — 3% Menthol
  Arms: Diclofenac Sodium/Menthol Gel; Menthol Gel
Drug: 0.09% Menthol — 0.09% Menthol
  Arms: Diclofenac Gel; Placebo Gel
Drug: 0.2% Sodium Lauryl Sulfate — 0.2% Sodium Lauryl Sulfate
  Arms: Sodium lauryl sulfate
Drug: 0.9% Saline — 0.9% Saline
  Arms: Saline

SUMMARY:
This research study is being conducted to investigate the skin irritancy potential of a new medication which contains two active ingredients (diclofenac and menthol) together in a gel formulation and is being developed to treat mild to moderate pain and inflammation, such as acute sport injuries, sprains and strains.

DETAILED DESCRIPTION:
Approximately 36 healthy subject volunteers will be exposed to seven test products (study treatment gel and six control products) simultaneously for 21 consecutive days. The seven test products will be applied using a 7-channel patch assembly that will be affixed to the infrascapular areas of the back of each subject for approximately 24 hours daily.

The subject will return to the clinic to undergo a skin irritation assessment at approximately 24 hours after the time the patch assembly was initially affixed.

During the visits, doctors or trained staff members will examine the signs of irritation (if any) of the skin where the test products are applied. The skin irritation assessment will primarily characterize the test products individually in terms of symptomatology using a 7-point categorical scale ranging from 1 (glazing and/or wrinkling) to 7 (erosion and/or vesiculation).

ELIGIBILITY:
Inclusion Criteria:

* Male/female volunteer ≥18 years
* No systemic/dermatologic disorder

Exclusion Criteria:

* Visible skin disease at the site of application that might interfere with skin assessments
* Allergy or hypersensitivity to NSAIDs or menthol or any of the excipients in the test product
* History of physical or psychiatric illness, or medical disorder
* Recent history of alcohol or drug abuse
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
Treatment mean cumulative irritation score | Day 21
  Cumulative irritation scores will be defined daily as the sum of irritation score and grade number
Adverse event assessment | 21 days + 5 days follow-up
  Adverse events will be graded on a three-point scale: 1. Mild-easily tolerated, causing minimal discomfort and not interfering with normal everyday activities; 2. Moderate-sufficiently discomforting to interfere with normal everyday activities; 3. Severe-any event that prevents normal everyday activities

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- TKL Research Inc, Paramus, New Jersey, United States

REFERENCES:
- See also: Results for the study 202187 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/202187?search=study&search_terms=202187#rs